CLINICAL TRIAL: NCT03971968
Title: Observational Study for the Long-Term Effects of a Dermal Substitute on Patients With Facial Burns.
Status: Completed | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Organisation for Burns, Scar Aftercare and Research (Other)
Responsible Party: Principal Investigator, Yamina Dupont, Medical Doctor, Universitair Ziekenhuis Brussel
Other Study IDs: CIP0019-201805-INT
Record Dates: First submitted 2019-05-23; First posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Cicatrix
Keywords: Burn; Scar; Face; Observational Study; Integra Artificial Skin
MeSH Terms: conditions — Cicatrix; Burns; Facies | interventions — Skin, Artificial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 = Intervention group: Group 1 suffered from third degree full thickness burns in the face/neck and received a surgical procedure with Integra Artificial Skin in the past
  Interventions: Procedure: Skin replacement with artificial skin
- Group 2 = Control Group: Group 2 is the healthy skin of a comparable and/or contralateral skin-site of the face/neck

INTERVENTIONS:
Procedure: Skin replacement with artificial skin — Integra® Dermal Regeneration Template is a bilayer membrane system for skin replacement. The dermal replacement layer is made of a porous matrix of fibers of cross-linked bovine tendon collagen and glycosaminoglycan (chondroitin-6-sulfate). The epidermal substitute layer is made of thin polysiloxane (silicone) layer to control moisture loss from the wound. The silicone outer layer temporarily closes the wound to ward off infection and control fluid and heat loss. As skin cells migrate into the matrix the collagen is slowly absorbed into the body and replaced with protein that is naturally produced by the skin. In approximately 14 to 21 days, new dermal skin is produced and the silicone layer can be removed. A thin skin graft of the person's epidermis is applied to the wound area to complete the procedure. In total, the two surgical procedures are typically completed within 30 days. A person is left with flexible growing skin and minimal damage at the skin graft donor sites.
  Other Names: Skin replacement with Integra Dermal Regeneration Template®
  Groups: Group 1 = Intervention group

SUMMARY:
The aim of this observational study is to investigate the long-term (between 10-20 years) results for the surgical treatment of third degree burn injury in the face and/or the neck by means of Integra® Dermal Regeneration Template.

This study is an observational case-control study. The healthy skin of a comparable and/or contralateral skin-site of the face/neck serves as a comparator.

The population consists of human volunteers between 18 and 75 years old with third degree full thickness burn injuries in the face and/or neck, who underwent surgical treatment with IDRT between 1998 and 2008.

DETAILED DESCRIPTION:
Study Procedures

Description of the clinical-investigation-related procedures in order of occurrence.

All patients will respect a 30 minute acclimatisation period in the measurement room with standardised room temperature (20-22°C) and relative humidity (40-50%). Patients will be asked to remove their silicones and pressure garments the evening before the actual measurement. The scar site used for testing is marked with a circular adhesive marking with a diameter of 30 mm. A picture is taken to establish the location. The following optimal patient positions are recommended. The patient is lying on his back with the arms next to the body.

Order of occurrence:

1. Intake questionnaire
2. Digital photographs and video recording
3. Patient and Observer Scar Assessment
4. Colour measurement
5. TEWL measurement
6. Elasticity measurement
7. Thickness measurement
8. Quality of Life questionnaires

Intake Questionnaire

Patient will be asked to fill out an intake form with all relevant information for the study. This will include age, body weight, gender, ethnicity, date of surgery, smoking, scar revision or initial treatment,

Digital Photographs and Video Recording

A digital photograph will be taken from the patient's face and/or neck. This photograph will be taken from a standardised distance. A video recording will be made to capture the mimic of the patient.

Patient and Observer reported Scar Assessment Scale (PSAS-OSAS)

The POSAS aims to measure scar quality. Current developments in scar treatment necessitate reliable and valid scar assessment tools. The POSAS is a comprehensive scale that is designed for the evaluation of all types of scars by professionals and patients. The Patient Scale gives the POSAS an important extra dimension because the patient's opinion is mandatory for a complete scar evaluation. When patients indicated may update their opinion without having to visit the hospital. This can be achieved at their convenience by internet or e-mail.

Clinimetric studies support the use of the POSAS for subjective scar evaluation. The first publication on the POSAS (Version 1.0) was in 2004. With one extra item for the Observer Scale and minor textual modifications POSASv2.0 was tested on linear scars and published in 2005.

The POSASv2.0 consists of two parts: a Patient Scale and an Observer Scale. Both scales contain six items that are scored numerically on a ten-step scale from 1 (= healthy skin) to 10 (= worst imaginable scar). Together they make up the 'Total Sum of Scores' of the Patient and Observer Scale. Furthermore category boxes are available to score nominal parameters (e.g. type of colour). Moreover, the patient and observer also score their 'Overall Opinion'.

Colour measurement with Mexameter® (Courage & Khazaka GmbH, Cologne, Germany)

Light is generated by a source lamp and is dispersed into its constituent wavelengths in a monochromator which results in a narrow band of the dispersed spectrum passing from the exit slit of the device. Suitable optics is used to lead this light, of a narrow wavelength band, to the sample being measured. A sample with an UV/Visible chromophore sample absorbs a certain amount of light and a suitable detector in the spectrophotometer detects the remaining light. The Beer-Lambert law is then applied to determine the concentration of the remaining light in the sample at a specific wavelength. The most commonly used wavelengths are 568 nm (green), 660 nm (red) and 880 nm (infrared). A melanin index can be computed from the results of red and infrared wavelengths and an erythema index is calculated from the results of green and red wavelengths.

TEWL measurements with Tewameter TM300® (Courage & Khazaka GmbH, Cologne, Germany)

The Tewameter® TEWL-probe is an open chamber system that measures water vapor permeability according to the diffusion principle. A probe, consisting of an open hollow cylinder of 20mm height and 10mm diameter measures the water evaporation gradient. Two sets of humidity and temperature sensors are placed in a measurement chamber at different heights above the scar/skin surface. At both points the local relative humidity and temperature are measured and the corresponding vapor pressure is calculated. The difference between the vapor pressure at both points is directly related to the rate of evaporative water loss. Results are expressed in g/m2/h.

Elasticity measurements with Cutometer® MPA580 (Courage & Khazaka Gmbh, Köln, Germany)

The Cutometer® is designed to measure elasticity of the upper skin layer using negative pressure which mechanically deforms the skin. The measuring principle is based on the suction method. Negative pressure is created in the device and the skin is drawn into the aperture of the probe and released again after a defined time. Inside the probe the penetration depth is determined by a non-contact optical measuring system. This optical measuring system consists of a light source and a light receptor and two prisms facing each other that project the light from transmitter to receptor. The light intensity varies due to the penetration depth of the skin. The resistance of the skin to the negative pressure (firmness) and its ability to return to its original position (elasticity) are displayed as curves (penetration depth in mm/time) in real time during the measurement. This measurement principle allows data collection on the elastic and mechanical properties of skin surface and enables objective quantification of skin aging. The Cutometer® measures the vertical deformation of the skin in millimetres when the skin is pulled by means of a controlled vacuum into the circular aperture of the probe.

Thickness measurement with DUB®Cutis High Frequency Ultrasound (Taberna Pro Medicum, Lüneberg, Germany)

The DUB®Cutis skinscanner is a 22-MHz frequency ultrasound scanning system with 57 µm resolution, a measuring depth of 10 mm and a 12,8 mm scan width. The system displays the information obtained in the form of a B-scan as either a colour or gray-scale image. The DUB system is an open system, preferably used with deionized water poured into the transducer through a special hole. To avoid leaking the user has to press the probe to the skin during the filling and the scanning procedure.

The result of ultrasonic imaging is usually presented in the form of A-scan (measurement at one point, showing the thickness of different layers of the skin), B-scan two-dimensional (2D) (cross-sectional view of the skin) and C-scan (2D) (view at some depth parallel to the surface of the skin) images.

EQ5D Quality of Life Questionnaire

The EQ-5D was developed by the EuroQol Group, an international, cross-disciplinary group that was set up in 1987 to investigate issues related to the evaluation of health. It has been translated to more than 60 languages, is used worldwide and has previously been used in Swedish populations. The reliability and validity of EQ-5D have been documented, both in general and in burns-specific populations.

The EQ-5D descriptive system encompasses five questions covering five dimensions: mobility, self-care, usual activities, pain and anxiety/depression. For each dimension, respondents value their health by reporting whether they are experiencing 1 = ''none'', 2 = ''moderate'' or 3 = ''extreme problems''. A unique EQ-5D health state is defined by combining the responses (1, 2 or 3) on each of the five dimensions. The EQ VAS is a vertical 20-cm line graded from 0 = ''worst possible health state'' to 100 = ''best possible health state'', on which the respondent is asked to mark his or her own current state of health. The EQ-5D health state can also be converted into a weighted index. The conversion into the index is based on norm values obtained in population-based enquiries. The EQ-5D index ranges from 0.594 = ''death or worse than death'' to 1 = ''full health''.

SF-36 Quality of Life Questionnaire

In development since the late 1980s, the SF-36 is a generic, psychometrically based, self-rated questionnaire. No less than five versions are available for use though the second (V2) and most recent format is the recommended option. It maps closely to the ICF domains and has published gender and age stratified norms for grouped, condition specific and individual comparisons. The SF-36 describes outcomes in terms of 8 separate subscales (domains) and three summary measures incorporating the domain scores. The survey may be administered in the standard or acute forms requesting responses in terms of recall of activity or feelings in the previous 4 weeks or 1 week, respectively. The reliability and validity of the SF-36 have been documented, both in general and in burns-specific populations.

Burn Specific Health Scale Brief (BSHS-B) Quality of Life Questionnaire

It is the only condition-specific health status instrument to be employed in patients with burns. This questionnaire was designed to assess the level of functioning and health-related QOL in adult burn survivors. The brief version (BSHS-B) was produced by Kildal et al. The BSHS-B has 40 items covering nine well-defined domains. Responses are rated on a 5-point scale from 0 (extremely) to 4 (none/not at all) for each of the 40 items and patients were asked to select the best answer. Mean scores are calculated for each of the domains. This final score reflects an alteration of the QOL. A higher mean score indicates a more positive evaluation of function and higher QOL.

ELIGIBILITY:
Inclusion Criteria:

* The subjects must be between 18 and 75 years old.
* Third degree full thickness burn injuries in the face and/or neck
* Having received surgical treatment with IDRT.
* Underwent surgery between 1998 and 2008.

Exclusion Criteria:

* Subjects with no matching control site comparable with assessed body location.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The population consists of human volunteers with third degree full thickness burn injuries in the face and/or neck, who underwent surgical treatment with IDRT.
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2019-02-14 (Actual)

PRIMARY OUTCOMES:
POSAS Patient Scale Total Sum of Scores | at enrolment
  The POSAS Patient Scale contains six items (pain, itch, colour, thickness, pliability, texture) that are scored numerically on a ten-step scale from 1 (= healthy skin) to 10 (= worst imaginable scar). Together they make up the 'Total Sum of Scores'.

SECONDARY OUTCOMES:
POSAS Observer Scale Total Sum of Scores | at enrolment
  The POSAS Observer Scale contains six items (vascularity, pigmentation, thickness, pliability, surface, texture) that are scored numerically on a ten-step scale from 1 (= healthy skin) to 10 (= worst imaginable scar). Together they make up the 'Total Sum of Scores'.
Objective colour measurements with Mexameter | at enrolment
  Mexameter is an objective assessment tool to measure erythema and pigmentation of the skin.
Objective thickness measurements with High Frequency Ultrasound | at enrolment
  With High Frequency Ultrasound one can measure the thickness of the dermis in µm.
Objective elasticity measurements with Cutometer | at enrolment
  Elasticity is measured objectively by means of skin suction.
Objective TEWL measurements with Tewameter | at enrolment
  The Tewameter measures the evaporation of water from the skin.
Quality of Life Questionnaire EQ5D | at enrolment
  This questionnaire assesses the mental and physical health and their consequences on quality of life. It is a generic questionnaire.
Quality of Life Questionnaire SF-36 | at enrollment
  This questionnaire assesses the mental and physical health and their consequences on quality of life. It is a generic questionnaire.
Quality of Life Questionnaire BSHS-B | at enrollment
  This questionnaire assesses the mental and physical health and their consequences on quality of life. It is a disease-specific questionnaire for patients with burn injuries.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Astrid Military Hospital, Neder-Over-Heembeek, Belgium